CLINICAL TRIAL: NCT02185274
Title: Observational Study on the Short- and Long-term Effects of Cross-sex-hormone Treatment on Metabolism and Psychopathology in Transsexuals Patients.
Brief Title: Observational Study on Metabolism and Psychopathology in Transsexual Patients
Status: Completed | Type: Observational
Sponsor: Max-Planck-Institute of Psychiatry (Other)
Collaborators: University of Erlangen-Nürnberg Medical School (Other); Institute for Sex Research and Forensic Psychiatry, Hamburg, Germany (Unknown); Hormon-und Stoffwechselzentrum München, Munich, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: MPIP-ENDO1
Record Dates: First submitted 2014-06-18; First posted 2014-07-09 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Transsexualism
Keywords: Transsexualism; Cross-sex hormone treatment; Sex hormones; Mood; Stress; Cortisol; Cardiovascular; Metabolome
MeSH Terms: conditions — Transsexualism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * 2 x 10ml serum
  * 10ml urine
  * Hair sample
  * 7,5ml EDTA-Blood for DNA and plasma
  * 2,5ml blood for mRNA-Analysis
  * 8,5ml stabilized serum
  * Stool sample (2-5ml)
Oversight: Data Monitoring Committee: No

SUMMARY:
Gender identity disorders (also known as transsexualism) is defined as a condition in which a person with apparently normal somatic sexual differentiation is convinced that he or she is actually a member of the other sex. Most patients therefore undergo so called cross-sex hormone treatment. Treatment protocols follow international consensus statements but vary considerably between different centres and countries since no prospective and controlled trials are available on this subject and recommendations are mainly based on retrospective data analysis and experience of the individual centres. Applying high doses of testosterone to biological females and vice versa high doses of estradiol to biological males definitely impacts myriads of body functions, from which it has to be assumed that only a minority has already been elucidated so far. Especially in male-to-female-transsexuals there seems to be an increased risk for the development of mood disorders and cardiometabolic comorbidities. In this multi-center observational study we want to investigate, if there is any difference with regard to these outcomes, according to the varying standards of cross-sex hormone treatment between the different centers. Different outcome measures described below will be assessed each time during routine visits at the different centers.

ELIGIBILITY:
Inclusion criteria

* Patients with the diagnosis gender identity disorder (ICD-10: F64.0), who have given written informed consent following adequate oral and written information.

General Exclusion criteria

* Patients below the age of 18
* Legally incompetent patients
* Prior intake of cross-sex hormones
* Missing written informed consent
* Intersexuality

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the outpatient clinics of the corresponding centres. Every patient is eligible who has not yet received any cross-sex hormone treatment. Patients will be invited to participate at the regular visit after which it is planned to start hormone treatment. Further visits will follow the regular check-up visits in the corresponding centers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-10; Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of depressive and anxious symptoms following initiation of cross-sex hormone treatment | Up to 5 years
  Incidence of depressive and anxious symptoms by means of clinical interview and questionnaires in the the study period defined by different cut-off points in the point scales of the corresponding questionnaire (Beck Depression Inventory II = BDII and Symptomcheckliste bei psychischen Störungen = SCL90 for depression and State and Trait Anxiety Inventory = STAI-X1, X2 for anxiety). A comparison will then be done between the different treatment modes.
Differences in the effects of the different treatment types on cardiometabolic parameters | Up to 5 years
  Differences in the effects of the different treatment types (differing in dose, application route and type of antiandrogen used) on cardiometabolic risk-parameters such as BMI, body-composition, fasting Insulin, fasting glucose, triglycerides, cholesterol, intima media thickness.

SECONDARY OUTCOMES:
Effects of cross-sex hormone treatment on cortisol secretion by hair cortisol measurements | Up to 5 years
  Assessment of cortisol secretion by a hair sample which provides information about the mean cortisol secretion during the last months. One cm of scalp hair resembles approximately 1 month of growth. This may provide additional information concerning overall cortisol secretion during the last 3 months. One small hair will be sampled by scalp and this will be analysed in regard to psychological and metabolic profiles.
Effects of cross-sex hormone treatment on stress-response by means of Dex/CRH-testing | Up to 5 years
  The Dex/CRH-Test has been in use for several years for testing the physiological cortisol-response in psychiatric and neurologic patients and is performed on a routine basis in the Max-Planck Institute for Psychiatry in patients suffering from depressive disorders. It is assumed that regulation of cortisol secretion and responsiveness of the hypothalamus-pituitary-adrenal (HPA)-axis is pathophysiologically related to depression. The test has been proven to be save. Common transient side-effects include flushing, palpitation, tachypnoea and feeling of warmth which usually resolve within minutes without further intervention.
Genetic predictors for treatment response | Up to 5 years
  Predictive value of different polymorphism in genes such as the ERa, ERb and AR (Androgen Receptor), GR (Glucocorticoid-Receptor) or genes involved in steroid metabolism and function on metabolic profiles, breast development and psychiatric outcome.
Effects of cross-sex hormone treatment on the metabolome | Up to 5 years
  Differences in plasma and urine metabolome in plasma such as amino acids; carbohydrates and related; catecholamines and related; complex lipids and related; energy metabolism and organic acids; fatty acids (free and from lipids); purines, pyrimidines and related; steroids and related; vitamins, cofactors and related.
Effects of cross-sex hormone treatment on peripheral neurotrophins | Up to 5 years
  Effects of cross-sex hormone treatment on serum Brain-Derived Neurotrophic Factor (BDNF) levels will be assessed in regular intervals during routine visits.
Association of hair cortisol and cortisol response during dex/crh-testing with psychopathology-scores assessed by clinical interview and questionnaires | Up to 5 years
  The following interviews will be used:
  * The MINI-PLUS interview assessing DSM axis I disorders [57].
  * The SCID-II interview assessing DSM axis II disorders
  The following questionaires will be used
  • stress coping (SVF-78)
  Personality:
  * personality (EPQ, TPQ,NEO-FFI)
  * self-reported quality of life (SF-36)
  * subjective body experience (FBeK)
  * self concept (SKI)
  * social support (B-Lor, FSOZ-U)
  * early life trauma (CTQ)
  Psychopathology:
  * State-Trait Anxiety Inventory (STAI Form X1, STAI Form X2)
  * Depressive symptoms (BDI II)
  * Psychopathology in general (SCL-90)
  Associations of cortisol- and ACTH response following dex/crg-challenge will be analyzed with regard to the presence of depression assessed by clinical interview and psychopathology scores assessed by BDI and STAIX. The other questionnaires will be used for multidimensional modelling.
Predictive value of hair cortisol and cortisol response in dex/crh-testing treatment for depression and anxiety | Up to 5 years
  Predictive value of hair cortisol 3 month at baseline and after treatment initiation and cortisol response at baseline and after 3 month after treatment initiation during dex/crh-testing for 12 month incidence of depressive or anxiety disorders assessed by clinical interview and questionnaires.
  The following interviews will be used:
  * The MINI-PLUS interview assessing DSM axis I disorders [57].
  * The SCID-II interview assessing DSM axis II disorders
  The following questionaires will be used
  * State-Trait Anxiety Inventory (STAI Form X1, STAI Form X2)
  * Depressive symptoms (BDI II)
  * Psychopathology in general (SCL-90)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias K Auer, MD, Principal Investigator — Max Planck Insitute of Psychiatry, Department of Neuroendocrinology
Locations (3):
- Germany (3):
  - Gynaecological department of the University hospital of Erlangen, Erlangen
  - Institute for Sex Research and Forensic Psychiatry, Hamburg
  - Hormon- und Stoffwechselzentrum München, Munich

REFERENCES:
- [Derived] Liwinski T, Auer MK, Schroder J, Pieknik I, Casar C, Schwinge D, Henze L, Stalla GK, Lang UE, von Klitzing A, Briken P, Hildebrandt T, Desbuleux JC, Biedermann SV, Holterhus PM, Bang C, Schramm C, Fuss J. Gender-affirming hormonal therapy induces a gender-concordant fecal metagenome transition in transgender individuals. BMC Med. 2024 Sep 2;22(1):346. doi: 10.1186/s12916-024-03548-z. PMID 39218875